CLINICAL TRIAL: NCT06245369
Title: Self-monitoring With Internet Technology to Choose Healthy Diets Study
Brief Title: SWITCH Diets Study: Self-monitoring With Internet Technology to Choose Healthy Diets
Acronym: SWITCH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Responsible Party: Principal Investigator, Brie Turner-McGrievy, Professor, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Pro00132921
Record Dates: First submitted 2024-01-29; First posted 2024-02-07 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Overweight and Obesity; Pre-diabetes
Keywords: Healthy diet, obesity, mobile technology, self-monitoring
MeSH Terms: conditions — Overweight; Obesity; Glucose Intolerance

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SWITCH tracking healthy nutrients (Experimental): Participants allocated to this group will be given goals to reach a recommended daily intake of nutrients in which US adults tend to not consume enough. Recommended amounts will be based off of age and sex, in line with the US Dietary Guidelines.
  Interventions: Behavioral: learning modules (within app); Behavioral: SWITCH app (self-regulation features) - Experimental
- standard SWITCH app (Active Comparator): Participants in this group will be given goals to reduce intake of nutrients in which US adults tend to consume too much. Personalized daily intake goals for nutrients will be based on age, weight, sex, and the US Dietary Guidelines.
  Interventions: Behavioral: learning modules (within app); Behavioral: SWITCH app (self-regulation features) - Comparator

INTERVENTIONS:
Behavioral: learning modules (within app) — Behavioral:
  Participants will have access to a weekly learning module created as Kahoot courses. Each module will include some or all (as applicable) of the following:
  * A brief educational video discussing the week's topic
  * A brief video sharing ideas for applying the educational content into daily life
  * PDF of "meal swap" examples
  * A weekly goal or challenge
  * Recipes
Behavioral: SWITCH app (self-regulation features) - Experimental — Behavioral:
  Diet (track by in app database). App homepage displays dietary intake graph -circles -. Participants will see an empty circles for the goal nutrients at the start of each day, which will fill up as the participant tracks his/her food intake. If the participant consumes an excess beyond the nutrient intake goal, the circle will remain entirely full.
  Arms: SWITCH tracking healthy nutrients
Behavioral: SWITCH app (self-regulation features) - Comparator — Diet (track by in app database). App homepage displays dietary intake graph -circles -.
  Participants allocated to the control group, tracking intake of nutrients to lower, will see a full circle at the start of each day which depletes, or empties, as the participant tracks his/her food intake. If the participant consumes an excess beyond the nutrient intake goal, the circle will remain entirely empty and the reported totals below the intake circles will display the current intake totals.
  Arms: standard SWITCH app

SUMMARY:
The goal of the Self-monitoring With Internet Technology to Choose Healthy Diets (SWITCH) study is to examine a 12-week remotely delivered program designed to help adults adopt a healthy dietary lifestyle and lose weight in a diverse cohort of adults with overweight/obesity.

The intervention uses a self-determination theory framework to provide a deeper understanding of the factors that influence dietary behavior within the context of tracking. This study incorporates autonomy-supportive strategies to encourage participants to feel more in control of their dietary choices and will provide information and resources to boost participant's competence in achieving their dietary goals. The intervention includes weekly learning modules to support healthy eating and weight loss and daily dietary tracking with visual feedback, all accessible within the SWITCH app.

DETAILED DESCRIPTION:
The SWITCH study is a 12-week remotely delivered, randomized behavioral intervention. Participants will be randomized to one of two groups: 1) SWITCH tracking nutrients to decrease (n=50) or 2) SWITCH tracking nutrients to increase (n=50). Participants will attend a study orientation, complete all baseline measures, be randomized, and then attend a training session for their group. In addition, participants will complete assessment at baseline and 12 weeks.

Intervention Design:

Diet tracking. Participants in both groups will be asked to track all meals, snacks, and beverages via the SWITCH app and complete a weekly learning module. Both groups will receive the same intervention, but the targeted nutrient goals and the in-app display of daily intake will differ between groups. Participants will be given goals to either increase certain nutrients or to decrease certain nutrients.

Diet related education to support healthy eating and weight loss will be provided each week within the SWITCH app. Each module includes some or all (as applicable) of the following components: A brief educational video discussing the week's topic, a video sharing ideas for applying the educational content into daily life, "meal swap" examples, a weekly goal or challenge and example recipes.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 64 years.
* BMI between 25 - 49.9 kg/m2
* Have 2 risk factors for T2DM in addition to having overweight or obesity (as defined by the NIDDK).
* Own and use a smartphone with a data plan.
* Must be willing and able to change dietary intake.
* Be free of major health or psychiatric diseases, drug, or alcohol dependency.
* Willing to sign informed consent.
* Own a digital body weight scale, have regular access, or be willing to purchase one

Exclusion Criteria:

* Currently participating in a weight loss program
* Has lost more than 10 pounds in the past 6 months.
* Diagnosed with type 2 diabetes or currently using medications that may impact blood glucose.
* Pregnant (or have been pregnant in the last 6 months), anticipating becoming pregnant in the next 12 months, or currently breastfeeding.
* Having an eating disorder.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2024-04-15 (Actual); Primary Completion 2025-02-14 (Actual); Study Completion 2025-03-18 (Actual)

PRIMARY OUTCOMES:
Change in Healthy Eating Index | 12 weeks
  Change in Healthy Eating Index from baseline to 12 weeks as assessed by dietary recalls.

SECONDARY OUTCOMES:
Change in Body weight | 12 weeks
  Change in Body weight assessed by home scale - self-report data confirmed by photo

CONTACTS AND LOCATIONS:
Overall Officials: Brie Turner-McGrievy, PhD, Principal Investigator — University of South Carolina
Locations (1):
- Prevention Research Center, University of South Carolina, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF